CLINICAL TRIAL: NCT05194670
Title: Comparison Between Bilateral Extended Depth of Focus (EDOF) Intraocular Lens Myopic Monovision and Monofocal Intraocular Lens Myopic Monovision for Myopic Patients: a Randomised Trial
Brief Title: Myopic Monovision: EDOF vs. Monofocal IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Myopic Monovision
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: Cataract; Myopia; enhanced depth of focus intraocular lens; mini-monovision
MeSH Terms: conditions — Cataract; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acunex Vario AN6V (Experimental): Patient will receive the enhanced depth of focus IOL during cataract surgery
  Interventions: Device: enhanced depth of focus IOL
- Acunex AN6 (Experimental): Patient will receive the monofocal IOL during cataract surgery
  Interventions: Device: monofocal IOL

INTERVENTIONS:
Device: enhanced depth of focus IOL — Acunex Vario AN6V, enhanced depth of focus IOL
  Arms: Acunex Vario AN6V
Device: monofocal IOL — Acunex AN6, monofocal IOL
  Arms: Acunex AN6

SUMMARY:
Comparison of EDOF IOLs versus monofocal IOLs with mini-monovision concerning intermediate and near visual acuity.

DETAILED DESCRIPTION:
Spectacle independence is one of the main aims in modern cataract surgery. Although bilateral monofocal IOL implantation, aiming for emmetropia or low myopia, leads to high levels of patient satifsfaction in distance vision, spectacle dependence for reading and other near vision tasks is the usual result.

There are different techniques to reduce spectacle dependence, the most common one is the use of multifocal IOLs. However, a variable number of patients complain of problems, such as glare or haloes. It appears that multifocal IOL technology does lead to less satisfying results in patients with pre-operative myopia. These patients are used to very good near vision when taking off their spectacles. Many of these patients would prefer to keep their distance spectacles and ideally would like to function well at intermediate and near distance without glasses for e.g. reading and computer- or household work.

One option to enhance intermediate vision and to leave patients with good contrast sensitivity is the use of extended depth of focus (EDOF) IOLs. One example is the ACUNEX Vario AN6V with a near add of 1.50 D. In particular, this design provides improved vision at a distance of 66 cm and more. Additional key features of the low-add IOL include good contrast sensitivity for twilight vision, optimized depth of focus, and natural imaging quality and color sensitivity.

Another option to allow spectacle independence is (mini-)monovision. For some people, who are in need of intermediate and near reading vision most of the time, mini-monovision with one eye having intermediate (arms length) and one eye having near (reading) vision is a good option ("myopic monovision").

Hence, the aim of the study is to analyse intermediate and near vision outcomes in myopic patients with either EDOF IOLs or monofocal IOLs with mini-monovision.

124 eyes of 62 patients will be included into this study. According to randomization, 31 patients will receive the EDOF IOLs (Acunex Vario AN6V) bilaterally, whereas in the other 31 patients a monofocal IOL (Acunex AN6) with mini-monovision will be implanted bilaterally. Follow-Up visits will be 1 hour, 1 week, and 2 months after surgery. A slit lamp examination, autorefraction and subjective refraction as well as visual acuity testing, reading performance, stereo vision testing and defocus curve assessment will be performed at this visits.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract in both eyes
* bilateral cataract surgery
* motivated to be less spectacle dependent in the intermediate to near vision range
* expected CDVA of 0.8 snellen or better
* myopic patients with shorter eye having an axial length of at least 25.5 mm
* age 21 and older
* planned postoperative astigmatis lower than or 0.75 D
* written informed consent prior to recruitment

Exclusion Criteria:

* pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* retinitis pigmentosa
* chronic uveitis
* amblyopia
* pupil decentration > 0.8 mm, pupil size < 2.8 mm
* preceded retinal surgery
* preceded LASIK
* any ophthalmic abnormality that could compromise visual function or the measurements

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Spectacle independence | 24 months
  Spectacle independence will be assessed using a questionnaire and compared between patients with EDOF IOLs and patients with the monofocal IOL

SECONDARY OUTCOMES:
Visual acuity | 24 months
  Visual acuity will be assessed using ETDRS charts and will be compared between patients with the EDOF IOLs and patients with the monofocal IOLs
Reading speed | 24 months
  Reading speed will be analysed by using the Salzburg Reading Desk and will be compared between patients with the EDOF IOLs and patients with the monofocal IOLs
Stereo vision | 24 months
  Stereo vision will be analysed by using a 3D-computer program and will be compared between patients with the EDOF IOLs and patients with the monofocal IOLs

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No